CLINICAL TRIAL: NCT06587113
Title: Contributions of Attentional and Inhibitory Functioning to Saccadic Decisions
Brief Title: An Investigation of Attentional and Inhibitory Processes During Active Visual Search in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-1148; R15EY035056-01 (NIH)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Eye Movements; Attention; Executive Function
Keywords: Individual differences; Eye movements; Perception; Attention; Inhibition
MeSH Terms: conditions — Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: Basic Experimental Studies Involving Humans (BESH)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): This study examines eye movement behavior using eye-tracking technology. Healthy participants perform three different tasks, including a visual search task, a stop-signal task, and a useful field of view task. Behavioral performance and eye movements are recorded for all tasks.
  Interventions: Other: Visual tasks

INTERVENTIONS:
Other: Visual tasks — In the experiments, participants sit in front of a computer screen with their head in a chinrest to control for distance from the monitor and eye-tracking equipment. For the visual search task, participants will search for a visual target among distractors and make a response regarding its orientation. For the stop-signal task, participants will make an eye movement to a target that appears on the screen, except on trials where a visual signal appears indicating they should cancel this behavior. In the useful field of view task, participants will report the location of a briefly-presented and masked target, while also responding to the identify of a central target in some blocks.

SUMMARY:
The goal of this study is to investigate the finding that there are large individual differences in how participants move their eyes during active visual search. For example, some individuals tend to fixate, that is point their eyes steadily at a single location, for longer than other individuals before moving to another location. This experiment will use behavioral tasks to measure an individual's attentional and inhibitory functioning, and then see how each of these contributes to between-participant variability in eye movement behavior during visual search.

DETAILED DESCRIPTION:
To accomplish the goal of understanding the source of individual variability in eye movement patterns, each participant will complete three separate tasks. The first task will require participants to find a target and eye movements will be measured to assess individual differences in fixation duration and other types of eye movement behavior. A second task will evaluate attentional functioning over the visual field by requiring participants to detect briefly-presented targets using their peripheral vision. Finally, a third task will assess inhibitory functioning by having participants attempt to stop eye movements after they have been programmed.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old

Exclusion Criteria:

* Self-reported history of neurological illness
* Uncorrected vision problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
First fixation duration during visual search | During visual search task
  This measure is the average first fixation duration during the visual search task. Possible scores are a minimum of 50 ms with an undeterminable positive number of ms as a maximum. This measure indicates the duration of processing before the first eye movement decision.
Fixation count during visual search | During visual search task
  This measure is the count the average number of eye movements participants made per trial during the visual search task. Possible scores range from a minimum of 0 to approximately 40 eye movements, given the time available. This measure indicates the amount of active exploration of the display during search.
Stop signal reaction time | During inhibitory task
  Stop signal reaction time is a quantitative estimate of how long participants take to successfully inhibit a planned eye movement. Possible scores range from a minimum of 0 ms to a maximum of about 600 ms. Low scores indicate strong inhibitory ability and high scores indicate weak inhibitory ability.
Useful field of view thresholding | During attention task
  Performance in a thresholding task indicates participants ability to detect a briefly presented target among distractors with 80% accuracy. Contrast of the displays varies until performance meets achieved level. Possible scores range from 0 to 100% contrast. Lower contrast indicates better information accrual, while higher contrast indicates worse.
Useful field of view dual task performance | During attention task
  Performance in a dual task indicates participants ability to spread attention across the visual field. Possible scores range from 0 to 100% accuracy. Higher performance indicates better information accrual, while lower performance indicates worse.

SECONDARY OUTCOMES:
Average fixation duration during visual search | During the visual search task
  This measure is the average fixation duration across all fixations in a trial during the visual search task. Possible scores range from a minimum of 50 ms to approximately 500 ms. This measure indicates the average duration of processing before a saccadic decision is made.

CONTACTS AND LOCATIONS:
Overall Officials: Carly J Leonard, Phd, Principal Investigator — University of Colorado enver
Locations (1):
- University of Colorado Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual data and analysis code will be shared through the Open Science Foundation (OSF) website.
Time Frame: The individual participant data and analysis code will be shared at the time when the manuscript reporting these results is submitted for publication.
URL: https://osf.io/67nz4/